CLINICAL TRIAL: NCT05144217
Title: Impact of Different Silymarin Dosages to Decrease Drug-induced Elevated Liver Enzymes Compared to Placebo in a Prospective Controlled Dose Finding Phase IIb Trial
Brief Title: Impact of Silymarin Dosages to Decrease Drug-induced Elevated Liver Enzymes Compared to Placebo
Acronym: SILVER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prof. Dr. Frank Behrens (Other)
Collaborators: Bionorica SE (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Frank Behrens, Sponsor representative, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMP-2501-2019-2
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Drug-induced Liver Injury
Keywords: silymarin
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Intervention Model Description: prospective placebo-controlled dose-finding study
Who Masked: Participant
Masking Description: study medication and placebo are provided in identical blister
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 1 capsule twice per day
  Interventions: Drug: Placebo
- oral administration of 2x 140 mg per day (Active Comparator): 1 capsule twice per day
  Interventions: Drug: 2x 140 mg per day
- oral administration of 3x 280 mg per day (Active Comparator): 2 capsules three times a day
  Interventions: Drug: 3x 280 mg per day
- oral administration of 1x 1120 mg per day (Active Comparator): 8 capsules once per day
  Interventions: Drug: 1x 1120 mg

INTERVENTIONS:
Drug: Placebo — 1 capsule per day of placebo
  Arms: Placebo
Drug: 2x 140 mg per day — 2 capsule per day of silimarit
  Arms: oral administration of 2x 140 mg per day
Drug: 3x 280 mg per day — 3 capsule per day of silimarit
  Arms: oral administration of 3x 280 mg per day
Drug: 1x 1120 mg — 8 capsule per day of silimarit
  Arms: oral administration of 1x 1120 mg per day

SUMMARY:
In this clinical study silymarin will be administered in different dosages and compared to placebo in order to address if the liver protecting features of silymarin, measured by changes of liver enzyme concentration, can be improved in patients with drug-induced elevated liver enzymes or drug-induced hepatocellular liver injury with higher systemic bioavailabilities due to administration of higher oral dosages or administration of higher administration frequency over a 35-day treatment period.

DETAILED DESCRIPTION:
In clinical routine care, drug-induced elevation of liver enzymes occurs often in parallel to new treatment initiation, possibly leading to interruption of treatment strategies if liver enzyme elevation does not normalize within 2 to 4 weeks.

Liver injury from medications usually occurs within 6 months of drug initiation and typically within the first 1-4 weeks1. In general, drug-induced liver injury (DILI) is related to the class of drug, the quantity of drug consumed, the patient's age and sex, and such concurrent factors as diabetes mellitus, excessive alcohol intake, e.g. high caloric diet, which can lead to NAFLD/steatosis, or the use of other medications. Drugs administered in higher doses are more likely to cause liver injury, especially drugs that require extensive hepatic metabolism1. Different forms of drug-induced elevation of liver enzymes can be differentiated according to localisation of the injury: hepatocellular or cholestatic liver injury or a mixture of both.Besides methotrexate and isozid, other medications have been reported to induce hepatocellular liver injury: acarbose, allopurinol, amiodarone, baclofen, bupropion, fluoxetine, ketoconazole, lisinopril, losartan, non-steroidal anti-inflammatory drugs (NSAIDs), omeprazole, paracetamol, paroxetine, pyrazinamide, rifampicin, risperidone, sertraline, statins, tetracyclines, trazodone, and valproic acid. Silymarin containing oral preparations are widely used for their liver protecting characteristics. The milk thistle ingredient silibinin is registered for continuous intravenous administration in the case of acute liver intoxications such as consumption of amanita mushrooms. Although its mode of action is still not clear, the clinical therapeutic benefits in patients with liver diseases are documented.

Pharmacokinetics of silymarin after oral administration are well understood. Due to its poor solubility in aqueous media, absorption from the intestinal tract is generally limited. Silymarin's systemic bioavailability of marketed products is therefore rather low, also because of predominant first pass biliary elimination. Exact PK/PD relations of the compound have not been assessed so far.

Hence, in this clinical study silymarin will be administered in different dosages and compared to placebo in order to address the following question: Can liver protecting features of silymarin, measured by changes of liver enzyme concentration, be improved in patients with drug-induced elevated liver enzymes or drug-induced hepatocellular liver injury with higher systemic bioavailabilities due to administration of higher oral dosages or administration of higher administration frequency over a 35-day treatment period?

ELIGIBILITY:
Inclusion Criteria:

Evidence of hepatocellular drug-induced injury due to treatment*

* ALT/AP ratio ≥ 5 ((ALT level/ALT upper limit of normal (ULN))/(AP level/AP ULN)) OR Evidence of drug-induced elevation of liver-enzymes
* ALT > 40 U/L and ≤ 2 x ULN
* ALT (> 40 U/L) ≥ 2 weeks and ≤ 3 months 3. Documentation (within the last 4 weeks before screening) of exclusion of liver tissue damage using either ultrasonography of the liver or Fibroscan with results ≤ 7 kPa (fibrosis score of F0 to F1) 4. BMI ≥ 18 and ≤ 30 5. Liver enzyme elevation inducing medication stable for ≥ 8 weeks before screening in the discretion of the treating physician 6. Written informed consent, after having been informed about potential benefit and potential risks of the clinical trial 7. Willing and capable to understand informed consent and follow the protocol

Exclusion Criteria:

1. Use of silymarin within the last 6 months
2. Current intake and intake within the last 4 weeks of drugs that have been shown to induce cholestatic or mixed hepatocellular/cholestatic liver injury (inducing cholestatic liver injury: amoxicilline and clavulanic acid, anabolic steroids, chlorpromazine, clopidogrel, erythromycin, irbesartan, mirtazapine, estrogen, terbinafine; inducing mixed liver injury: amitriptyline, azathioprine, captopril, carbamazepine, clindamycin, co-trimoxazole, cyproheptadine, enalapril, flutamide, nitrofurantoin, phenobarbital, phenytoin, sulphonamide, trazodone, verapamil)
3. Patients with chronic liver disease, existing fibrosis or cirrhosis
4. Patients with acute viral hepatitis, autoimmune hepatitis or immune-mediated hepatitis (e.g., with immune checkpoint inhibitor treatment), acute Budd-Chiari syndrome, Wilson disease, and ischemic liver injury
5. Cholestatic or mixed hepatocellular/mixed liver injury
6. Patients with diabetes types 1 or 2
7. Any malignancy within the past 5 years
8. Patients with chronic intestinal diseases (e.g., ulcerative colitis) and intestinal barrier dysfunction in the discretion of the treating physician (e.g., patient can be included if disease is judged as stable by the treating physician with no likely interference with the study outcomes and the safety of the patient)
9. Evidence of significant uncontrolled concomitant diseases or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome
10. History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
11. Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations, e.g. milk thistle, soy oil, peanut (according to Summary of Product Characteristics (SmPc))
12. Contraindications to use the investigational medicinal product (IMP), e.g. hereditary galactose intolerance, genetic lactase deficiency or glucose-galactose malabsorption (according to SmPC)
13. Subjects with severe or moderate allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
14. Laboratory values other than target parameters out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
15. Positive anti-HIV-test, antiHBs- or anti-HCV-test at Screening
16. History of or current drug or alcohol dependence
17. Subjects with a positive drug test at screening (incl. alcohol)
18. Regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol for male or ≥ 20 g pure ethanol for female per day
19. Participation in a clinical trial during the last two months prior to individual enrolment of the subject or current participation
20. Use of drugs during the last two weeks prior Baseline that can affect absorption (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists)
21. Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial
22. Subjects who do not agree to apply adequate contraceptive methods as defined in Note for Guidance on Non-Clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (CPMP/ICH/286/95, modification), November 2000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in blood ALT (Alanine-Aminotransferase) in IU/L | at day 35
  Change in blood ALT in IU/Lin all treatment groups

SECONDARY OUTCOMES:
Liver enzyme blood parameter AST (Aspartate-Aminotransferase) | Baseline (prior treatment)
  Change of Liver enzyme blood parameter AST in IU/Lin all treatment groups
Liver enzyme blood parameter AST | Day 7
  Change of Liver enzyme blood parameter AST in IU/Lin all treatment groups
Liver enzyme blood parameter AST | Day 14
  Change of Liver enzyme blood parameter AST in IU/Lin all treatment groups
Liver enzyme blood parameters: AST | Day 21
  Change of Liver enzyme blood parameter AST in IU/Lin all treatment groups
Liver enzyme blood parameter AST | Day 28
  Change of Liver enzyme blood parameter AST in IU/Lin all treatment groups
Change Liver enzyme blood parameter AST | Day 35
  Change of Liver enzyme blood parameter AST in IU/Lin all treatment groups
Change Liver enzyme blood parameter ALT | Baseline
  Change of Liver enzyme blood parameter ALT in IU/Lin all treatment groups
Change Liver enzyme blood parameter ALT | Day 7
  Change of Liver enzyme blood parameter ALT in IU/Lin all treatment groups
Change Liver enzyme blood parameter ALT | Day 14
  Change of Liver enzyme blood parameter ALT in IU/Lin all treatment groups
Change Liver enzyme blood parameter ALT | Day 21
  Change of Liver enzyme blood parameter ALT in IU/Lin all treatment groups
Change Liver enzyme blood parameter ALT | Day 28
  Change of Liver enzyme blood parameter ALT in IU/Lin all treatment groups
Change Liver enzyme blood parameter ALT | Day 35
  Change of Liver enzyme blood parameter ALT in IU/Lin all treatment groups
Change Liver enzyme blood parameter GGT (Gamma-Glutamyl-Transferase) | Baseline
  Change of Liver enzyme blood parameter GGT in IU/Lin all treatment groups
Change Liver enzyme blood parameter GGT (Gamma-Glutamyl-Transferase) | Day 7
  Change of Liver enzyme blood parameter GGT in IU/Lin all treatment groups
Change Liver enzyme blood parameter GGT (Gamma-Glutamyl-Transferase) | Day 14
  Change of Liver enzyme blood parameter GGT in IU/Lin all treatment groups
Change Liver enzyme blood parameter GGT (Gamma-Glutamyl-Transferase) | Day 21
  Change of Liver enzyme blood parameter GGT in IU/Lin all treatment groups
Change Liver enzyme blood parameter GGT (Gamma-Glutamyl-Transferase) | Day 28
  Change of Liver enzyme blood parameter GGT in IU/Lin all treatment groups
Change Liver enzyme blood parameter GGT (Gamma-Glutamyl-Transferase) | Day 35
  Change of Liver enzyme blood parameter GGT in IU/Lin all treatment groups
Change Liver enzyme blood parameter AP (Alkaline phosphatase ) | Baseline
  Change of Liver enzyme blood parameter AP in IU/Lin all treatment groups
Change Liver enzyme blood parameter AP (Alkaline phosphatase ) | Day 7
  Change of Liver enzyme blood parameter AP in IU/Lin all treatment groups
Change Liver enzyme blood parameter AP (Alkaline phosphatase ) | Day 14
  Change of Liver enzyme blood parameter AP in IU/Lin all treatment groups
Change Liver enzyme blood parameter AP (Alkaline phosphatase ) | Day 21
  Change of Liver enzyme blood parameter AP in IU/Lin all treatment groups
Change Liver enzyme blood parameter AP (Alkaline phosphatase ) | Day 28
  Change of Liver enzyme blood parameter AP in IU/L in all treatment groups
Change Liver enzyme blood parameter AP (Alkaline phosphatase ) | Day 35
  Change of Liver enzyme blood parameter AP in IU/L in all treatment groups
Change Liver enzyme blood parameter bilirubin | Baseline
  Change of Liver enzyme blood parameter bilirubin in all treatment groups
Change Liver enzyme blood parameter bilirubin | Day 7
  Change of Liver enzyme blood parameter bilirubin in all treatment groups
Change Liver enzyme blood parameter bilirubin | Day 14
  Change of Liver enzyme blood parameter bilirubin in all treatment groups
Change Liver enzyme blood parameter bilirubin | Day 21
  Change of Liver enzyme blood parameter bilirubin in all treatment groups
Change Liver enzyme blood parameter bilirubin | Day 28
  Change of Liver enzyme blood parameter bilirubin in all treatment groups
Change Liver enzyme blood parameter bilirubin | Day 35
  Change of Liver enzyme blood parameter bilirubin in all treatment groups
Change Liver enzyme blood parameter INR (International Normalized Ratio) | baseline
  Change of Liver enzyme blood parameter INR in all treatment groups
Change Liver enzyme blood parameter INR (International Normalized Ratio) | Day 7
  Change of Liver enzyme blood parameter INR in all treatment groups
Change Liver enzyme blood parameter INR (International Normalized Ratio) | Day 14
  Change of Liver enzyme blood parameter INR in all treatment groups
Change Liver enzyme blood parameter INR (International Normalized Ratio) | Day 21
  Change of Liver enzyme blood parameter INR in all treatment groups
Change Liver enzyme blood parameter INR (International Normalized Ratio) | Day 28
  Change of Liver enzyme blood parameter INR in all treatment groups
Change Liver enzyme blood parameter INR (International Normalized Ratio) | Day 35
  Change of Liver enzyme blood parameter INR in all treatment groups
Change Liver enzyme blood parameter Quick value | baseline
  Change of Liver enzyme blood parameter Quick value in all treatment groups
Change Liver enzyme blood parameter Quick value | Day 7
  Change of Liver enzyme blood parameter Quick value in all treatment groups
Change Liver enzyme blood parameter Quick value | Day 14
  Change of Liver enzyme blood parameter Quick value in all treatment groups
Change Liver enzyme blood parameter Quick value | Day 21
  Change of Liver enzyme blood parameter Quick value in all treatment groups
Change Liver enzyme blood parameter Quick value | Day 28
  Change of Liver enzyme blood parameter Quick value in all treatment groups
Change Liver enzyme blood parameter Quick value | Day 35
  Change of Liver enzyme blood parameter Quick value in all treatment groups
Change ALT/AP ratio | baseline
  Change of ALT/AP ratio in all treatment groups
Change ALT/AP ratio | Day 7
  Change of ALT/AP ratio in all treatment groups
Change ALT/AP ratio | Day 14
  Change of ALT/AP ratio in all treatment groups
Change ALT/AP ratio | Day 21
  Change of ALT/AP ratio in all treatment groups
Change ALT/AP ratio | Day 28
  Change of ALT/AP ratio in all treatment groups
Change ALT/AP ratio | Day 35
  Change of ALT/AP ratio in all treatment groups
Lipids analysis | Baseline
  LDL (Low Density Lipoproteins) in all treatment groups
Lipids analysis LDL | Day 7
  LDL (Low Density Lipoproteins) in all treatment groups
Lipids analysis LDL | Day 14
  LDL (Low Density Lipoproteins) in all treatment groups
Lipids analysis LDL | Day 21
  LDL (Low Density Lipoproteins) in all treatment groups
Lipids analysis LDL | Day 28
  LDL (Low Density Lipoproteins) in all treatment groups
Lipids analysis LDL | Day 35
  LDL (Low Density Lipoproteins) in all treatment groups
Lipids analysis | baseline
  HDL (High Density Lipoproteins) in all treatment groups
Lipids analysis | Day 7
  HDL (High Density Lipoproteins) in all treatment groups
Lipids analysis | Day 14
  HDL (High Density Lipoproteins) in all treatment groups
Lipids analysis | Day 21
  HDL (High Density Lipoproteins) in all treatment groups
Lipids analysis | Day 28
  HDL (High Density Lipoproteins) in all treatment groups
Lipids analysis | Day 35
  HDL (High Density Lipoproteins) in all treatment groups
Lipids analysis | Day baseline
  VLDL (very low Density Lipoproteins) in all treatment groups
Lipids analysis VLDL | Day 7
  VLDL (very low Density Lipoproteins) in all treatment groups
Lipids analysis VLDL | Day 14
  VLDL (very low Density Lipoproteins) in all treatment groups
Lipids analysis VLDL | Day 21
  VLDL (very low Density Lipoproteins) in all treatment groups
Lipids analysis VLDL | Day 28
  VLDL (very low Density Lipoproteins) in all treatment groups
Lipids analysis VLDL | Day 35
  VLDL (very low Density Lipoproteins) in all treatment groups
Lipids analysis triglycerides | baseline
  triglycerides in all treatment groups
Lipids analysis triglycerides | Day 7
  triglycerides in all treatment groups
Lipids analysis triglycerides | Day 14
  triglycerides in all treatment groups
Lipids analysis triglycerides | Day 21
  triglycerides in all treatment groups
Lipids analysis triglycerides | Day 28
  triglycerides in all treatment groups
Lipids analysis triglycerides | Day 35
  triglycerides in all treatment groups
Lipids analysis total cholesterol | baseline
  total cholesterol in all treatment groups
Lipids analysis total cholesterol | Day 7
  total cholesterol in all treatment groups
Lipids analysis total cholesterol | Day 14
  total cholesterol in all treatment groups
Lipids analysis total cholesterol | Day 21
  total cholesterol in all treatment groups
Lipids analysis total cholesterol | Day 28
  total cholesterol in all treatment groups
Lipids analysis total cholesterol | Day 35
  total cholesterol in all treatment groups
bloodparameter assessment | baseline
  fasting glucose value in all treatment groups
bloodparameter assessment | Day 7
  fasting glucose value in all treatment groups
blood parameter assessment | Day 14
  fasting glucose value in all treatment groups
blood parameter assessment | Day 21
  fasting glucose value in all treatment groups
blood parameter assessment | Day 28
  fasting glucose value in all treatment groups
blood parameter assessment | Day 35
  fasting glucose value in all treatment groups
Proportion of patients with normalization in liver enzyme blood parameters | Day 35
  normalisation of liver enzyme blood parameters such as AST (< 40 IU/L), ALT (< 40 IU/L), GGT, AP, bilirubin, INR, Quick
Plasma silymarin dose concentration | Base line
  concentration of silymarin
Plasma silymarin dose concentration | day 7
  concentration of silymarin
Plasma silymarin dose concentration | day 14
  concentration of silymarin
Plasma silymarin dose concentration | day 21
  concentration of silymarin
Plasma silymarin dose concentration | day 28
  concentration of silymarin
Plasma silymarin dose concentration | day 35
  concentration of silymarin
Fibroscan value | baseline
  measurement of Fibroscan
Fibroscan value | day 14
  measurement of Fibroscan
Fibroscan value | day 35
  measurement of Fibroscan
Fibrosis score | baseline
  score F0 to F4
Fibrosis score | Day 14
  score F0 to F4
Fibrosis score | Day 35
  score F0 to F4
CAP score | baseline
  score measured in dB/m
CAP score | day 14
  score measured in dB/m
CAP score | day 35
  score measured in dB/m
Body Mass Index (BMI) | baseline
  index measured in weight and height
Silymarin concentration in blood plasma in pharmakokinetic substudy - AUC | baseline
  assessement of area under the curve (AUC),
Silymarin concentration in blood plasma in pharmakokinetic substudy - tmax | baseline
  assessement of time to maximal concentration (tmax)
Silymarin concentration in blood plasma in pharmakokinetic substudy - Cmax | baseline
  assessement of maximal concentration (Cmax)
Treatment adherence | Baseline
  measured by patient diary
Treatment adherence | Day 7
  measured by patient diary
Treatment adherence | Day 14
  measured by patient diary
Treatment adherence | Day 21
  measured by patient diary
Treatment adherence | Day 28
  measured by patient diary
Treatment adherence | Day 35
  measured by patient diary
quality of life measurements | baseline
  measured by short form survey (SF36) questionnaire
quality of life measurements | Day 7
  measured by short form survey (SF36) questionnaire
quality of life measurements | Day 14
  measured by short form survey (SF36) questionnaire
quality of life measurements | Day 21
  measured by short form survey (SF36) questionnaire
quality of life measurements | Day 28
  measured by short form survey (SF36) questionnaire
quality of life measurements | Day 35
  measured by short form survey (SF36) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Schaefer, MD, Study Chair — Fraunhofer ITMP
Locations (2):
- Germany (2):
  - Universtity Hospital - clinic for dermatology, venerology and allergology, Frankfurt, Hessia
  - CIRI, Frankfurt, Hessia

IPD SHARING:
Plan to Share IPD: No